CLINICAL TRIAL: NCT00393042
Title: Sleep and Tolerability of Extended Release Dexmethylphenidate vs. Mixed Amphetamine Salts: A Double Blind, Placebo Controlled Study (SAT STUDY)
Brief Title: Sleep and Tolerability Study: Comparing the Effects of Adderall XR and Focalin XR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Mark Stein, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRIT124E US15; 2006-0423; 2006-04
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; sleep; side effects; stimulants
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride; SLI381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Focalin XR then Adderall XR (Experimental): Subjects are given the Focalin XR first (dexmethylphenidate) for four weeks with a randomized placebo week followed by Adderall XR (mixed amphetamine salts) for four weeks with a randomized placebo week.
  Interventions: Drug: Dexmethylphenidate; Drug: Mixed Amphetamine Salts, ER; Drug: placebo
- Adderall XR then Focalin XR (Experimental): Subjects are given the Adderall XR (mixed amphetamine salts) for four weeks with a randomized placebo week followed by Focalin XR first (dexmethylphenidate) for four weeks with a randomized placebo week.
  Interventions: Drug: Dexmethylphenidate; Drug: Mixed Amphetamine Salts, ER; Drug: placebo

INTERVENTIONS:
Drug: Dexmethylphenidate — 10, 20, 25-30 mg.
  Other Names: Focalin XR
Drug: Mixed Amphetamine Salts, ER — 10, 20, 25-30
  Other Names: Adderall XR
Drug: placebo — randomized placebo week during each 4 week period

SUMMARY:
The purpose of this study is to evaluate how children and adolescents with Attention Deficit/ Hyperactivity Disorder (ADHD) respond to treatment with three differing doses of stimulant medications used to treat ADHD, Adderall XR® and Focalin XR®. Another purpose of the study is to evaluate if there are differences in sleep and other side effects, such as changes in mood or loss of appetite, which can occur with stimulant medications. A third purpose is to determine if there are differences in the characteristics of individuals who respond better to either of the medications.

This research is being done because the investigators do not know if one of these two commonly used treatments is better tolerated than the other. Children and adolescents with ADHD often have a hard time sitting still, playing quietly, finishing things they start, paying attention, waiting their turn, and not distracting others. These medications improve these symptoms, but sometimes affect sleep, appetite, or mood.

It is hypothesized that at effective and frequently prescribed doses, Adderall will be associated with insomnia, more stimulant side effects, and decreased tolerability during an acute trial relative to Focalin.

DETAILED DESCRIPTION:
ADHD is often treated with stimulant medications, which have demonstrated short-term efficacy in numerous trials. However, treatment is often discontinued prematurely. Although ADHD often persists through adolescence, approximately half of all children who are treated with a stimulant medication discontinue treatment within one year (Charach, Ickowicz et al. 2004). Presumably, tolerability and treatment compliance are highly related to the side effect profile of stimulant medications (Schachar, Jadad et al. 2002). Sleep problems, particularly insomnia, are frequently associated with ADHD and are often exacerbated by stimulant medications, particularly at higher doses. Other frequent stimulant side effects are decreased appetite and mood lability (dysphoria/euphoria). Little is known about the relative effects of different stimulant formulations and dosages (i.e amphetamine, methylphenidate, dexmethylphenidate) on sleep and tolerability. There is some preliminary data with short acting stimulants suggesting a higher prevalence of sleep and appetite problems with amphetamine relative to mph (Pelham, Aronoff et al. 1999). Several studies indicate that sleep and other stimulant side effects are dose related (Stein, Sarampote et al. 2003), although this has not been found in all studies. Moreover, it is unclear if there are differences between long-acting amphetamine and methylphenidate based stimulants in their side effect profile and tolerability. Thus, we will directly compare these two long acting stimulant medications on their side effect profile and tolerability, including measures of sleep, mood, and evening behavior (e.g., family conflicts). The recently developed extended release formulation of dexmethylphenidate will be compared to one of the most common treatments for ADHD, extended release formulation of mixed amphetamine salts. The subject population will be older children and adolescents (10-17) with ADHD who are most likely to be treated with moderate to higher dose levels of stimulant medications and can complete all self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Any ADHD subtype, determined by KSADS interview (Kaufman, Birmaher et al. 1997). Comorbidity will likewise be allowed, to ensure representation.
* Signed informed consent and assent
* Clinical Global Impressions - Severity for ADHD (CGI-S-ADHD) rating is greater than or equal to 4
* Findings on physical exam, laboratory studies, vital signs, and ECG are judged to be normal for age
* Pulse and blood pressure are within 95% of age and gender mean
* Able to complete study instruments and swallow capsules
* Willing to commit to the entire visit schedule for the study, including at least one visit to UIC Medical Center.

Exclusion Criteria:

* Previous diagnosis of mental retardation
* Non-responder to either medication at the doses offered in the study in an adequate trial
* Must not have experienced disabling adverse effects with either medication
* Concomitant psychotropic medications are required or medications which might have a CNS effect
* Any other medical condition which represents a contraindication for either treatment is present
* History of alcohol or drug abuse in the past 3 months, or a positive urinary toxic screen on initial evaluation that is not explained by a time-limited medical circumstance
* Females of childbearing age who are sexually active, do not use acceptable birth control (double protection method), and after counseling, are unwilling to do so
* History of allergic reactions to multiple medications
* A history of psychosis
* Diagnosis of bipolar disorder

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Stein, PhD, Principal Investigator — University of Illinois-Chicago; Hyperactivity, Attention and Learning Problems Clinic (HALP); Elizabeth Charney, MD, Principal Investigator — University of Illinois-Chicago, Hyperactivity, Attention, and Learning Problems Clinic (HALP)
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Northbrook HALP Clinic/ADHD Research Center, Northbrook, Illinois

REFERENCES:
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Charach A, Figueroa M, Chen S, Ickowicz A, Schachar R. Stimulant treatment over 5 years: effects on growth. J Am Acad Child Adolesc Psychiatry. 2006 Apr;45(4):415-21. doi: 10.1097/01.chi.0000199026.91699.20. PMID 16601646
- [Background] Schachar R, Jadad AR, Gauld M, Boyle M, Booker L, Snider A, Kim M, Cunningham C. Attention-deficit hyperactivity disorder: critical appraisal of extended treatment studies. Can J Psychiatry. 2002 May;47(4):337-48. doi: 10.1177/070674370204700404. PMID 12025432
- [Background] Pelham WE, Aronoff HR, Midlam JK, Shapiro CJ, Gnagy EM, Chronis AM, Onyango AN, Forehand G, Nguyen A, Waxmonsky J. A comparison of ritalin and adderall: efficacy and time-course in children with attention-deficit/hyperactivity disorder. Pediatrics. 1999 Apr;103(4):e43. doi: 10.1542/peds.103.4.e43. PMID 10103335
- [Background] Stein MA, Sarampote CS, Waldman ID, Robb AS, Conlon C, Pearl PL, Black DO, Seymour KE, Newcorn JH. A dose-response study of OROS methylphenidate in children with attention-deficit/hyperactivity disorder. Pediatrics. 2003 Nov;112(5):e404. doi: 10.1542/peds.112.5.e404. PMID 14595084
- [Result] Stein MA, Waldman ID, Charney E, Aryal S, Sable C, Gruber R, Newcorn JH. Dose effects and comparative effectiveness of extended release dexmethylphenidate and mixed amphetamine salts. J Child Adolesc Psychopharmacol. 2011 Dec;21(6):581-8. doi: 10.1089/cap.2011.0018. Epub 2011 Dec 2. PMID 22136094
- [Derived] Santisteban JA, Stein MA, Bergmame L, Gruber R. Effect of extended-release dexmethylphenidate and mixed amphetamine salts on sleep: a double-blind, randomized, crossover study in youth with attention-deficit hyperactivity disorder. CNS Drugs. 2014 Sep;28(9):825-33. doi: 10.1007/s40263-014-0181-3. PMID 25056567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from the investigators' practices, clinic referrals, and radio advertisements. Participants were enrolled between January 2007 and January 2009.
Pre-assignment Details: 7 participants didn't want to participate after screening, 1 didn't meet criteria, 1 ADHD was not the primary condition, 1 showed an abnormal lab/physical/EKG, 1 was unable to swallow pills, 1 had an exclusionary medical condition, 1 was removed due to protocol violations.
Groups:
- Focalin XR Then Adderall XR: Focalin XR first for 4 weeks (3 dose levels and placebo) then Adderall XR for 4 weeks (3 dose levels and placebo).
- Adderall XR Then Focalin XR: Adderall XR first for 4 weeks (3 dose levels and placebo) then Focalin XR for 4 weeks (3 dose levels and placebo).
Period: First Intervention
Arm/Group | Focalin XR Then Adderall XR | Adderall XR Then Focalin XR
Started | 31 | 33
Completed the Placebo Dosage | 27 | 29
Completed 10mg Dosage | 29 | 29
Completed 20 mg Dosage | 26 | 28
Completed 25/30mg Dosage | 27 | 27
Completed | 26 | 27
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervetion
Arm/Group | Focalin XR Then Adderall XR | Adderall XR Then Focalin XR
Started | 26 | 27
Completed Placebo Dosage | 25 | 21
Completed 10 mg Dosage | 26 | 24
Completed the 20mg Dosage | 24 | 21
Completed 25/30 mg Dosage | 24 | 20
Completed | 24 | 19
Not Completed | 2 | 8
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: 77 individuals were screened , 13 patients were excluded, 64 patients were randomized. Of the 64 randomized, 21 discontinued at various points during the trial.
Groups:
- Overall Study: Participants either Adderall XR or Focalin XR for four weeks (3 dose levels and placebo) followed by four weeks (3 dose levels and placebo) of the opposite medication they received the first four weeks. Baseline Measures are based off all participants that were randomized regardless of the order they received the medication. Since we were interested in evaluating efficacy and adverse events at all dose conditions, participants were included in analysis if they received at least 2 weeks of study drug to insure that all participants had been exposed to at least one week of active drug
Arm/Group | Overall Study
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (2.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Sleep Start Time, and End Time as Determined by Actigraph and Sleep Diary Over 8 Weeks.
Description: Actigraphs (AW64 series) were worn each night and were used to assess participant's sleep patterns in their natural home environment. These computerized wristwatch-like devices collect data generated by movements. They are minimally invasive and allow sleep to be recorded reliably without interfering with the family's routine. One-minute epochs were used to analyze actigraphic sleep sata. Bedtimes and wake times were reported for each participant using sleep logs, and these times were used as the start and end times for the analyses. For each 1-min epoch, the total sum of activity counts were computed. If they exceeded a threshold (threshold sensitivity value = mean score in active period/45), then the epoch was considered waking. If it fell below that threshold, then it was considered sleep. The data for Adderall XR and Focalin XR was combined to look at the cumulative effects that medication has on sleep.
Time Frame: 8-10 weeks
Population: Subjects with complete and valid actigraphy (n = 37) and sleep diaries were used to calculate sleep onset latency and sleep duration.
Measure: Mean (Standard Deviation); unit: HHMM.SS
Groups:
- Placebo: Regardless of the medication the participants were taking, each 4 week period included a randomized placebo week. This data is based off each participant's placebo weeks.
- 10mg of Either Focalin XR or Adderall XR: Each participant received 10mg of either Focalin XR or Adderall XR. The data collected from the 10mg week of both drugs was combined.
- 20mg of Either Focalin XR or Adderall XR: Each participant received 20mg of either Focalin XR or Adderall XR. The data collected from the 20mg week of both drugs was combined.
- 25/30mg of Either Focalin XR or Adderall XR: Each participant received 25 or 30mg of either Focalin XR or Adderall XR depending on their weight. The data collected from the 25/30mg week of both drugs was combined.
- Adderall XR All Dose Levels: Participants were given 10mg, 20mg, 25/30mg (depending on their weight) and a randomized placebo week for 4 weeks. This data is combines the 10mg, 20mg, and 25/30mg data for Adderall XR.
- Focalin XR All Dose Levels: Participants were given 10mg, 20mg, 25/30mg (depending on their weight) and a randomized placebo week for 4 weeks. This data is combines the 10mg, 20mg, and 25/30mg data for Focalin XR.
Arm/Group | Placebo | 10mg of Either Focalin XR or Adderall XR | 20mg of Either Focalin XR or Adderall XR | 25/30mg of Either Focalin XR or Adderall XR | Adderall XR All Dose Levels | Focalin XR All Dose Levels
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
HHMM.SS
  Sleep start time | 2249 (0012.19) | 2304 (0010.40) | 2319 (0012.21) | 2325 (0011.17) | 2309 (0011.05) | 2309 (0011.19)
  Sleep End time | 0742 (0015.36) | 0728 (0009.54) | 0735 (0010.46) | 0732 (0011.09) | 0735 (0010.40) | 0734 (0010.04)

2. Primary Outcome: Sleep Duration
Description: Actigraphs (AW64 series) were worn each night and were used to assess participant's sleep patterns in their natural home environment. These computerized wristwatch-like devices collect data generated by movements. They are minimally invasive and allow sleep to be recorded reliably without interfering with the family's routine. One-minute epochs were used to analyze actigraphic sleep sata. Bedtimes and wake times were reported for each participant using sleep logs, and these times were used as the start and end times for the analyses. For each 1-min epoch, the total sum of activity counts were computed. If they exceeded a threshold (threshold sensitivity value = mean score in active period/45), then the epoch was considered waking. If it fell below that threshold, then it was considered sleep.The data for Adderall XR and Focalin XR was combined to look at the cumulative effects that medication has on sleep.
Time Frame: 8-10 weeks
Population: participants with sufficient sleep actigraphy data for analysis (n=37)
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 20 mg of Either Focalin XR or Adderall XR: Each participant received 20mg of either Focalin XR or Adderall XR. The data collected from the 20mg week of both drugs was combined.
- 25/30mg of Either Focalin XR or Adderall XR: Each participant received 25/30mg of either Focalin XR or Adderall XR depending on their weight. The data collected from the 25/30mg week of both drugs was combined.
Arm/Group | Placebo | 10mg of Either Focalin XR or Adderall XR | 20 mg of Either Focalin XR or Adderall XR | 25/30mg of Either Focalin XR or Adderall XR | Adderall XR All Dose Levels | Focalin XR All Dose Levels
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37 | 37
minutes | 459.6 (73.6) | 446.7 (63.58) | 432.17 (64.6) | 425.5 (61.5) | 438.82 (67.2) | 443.2 (66.9)

3. Secondary Outcome: ADHD Parent Rating Scale-IV
Description: Measures the severity of Total ADHD symptoms, Inattention and Hyperactivity/Impulsive symptoms. The Inattention and Hyperactivity/Impulsive symptoms can range from 0 to 27 each, with a higher score reflecting more severe ADHD symptoms. The total score is calculated by summing the inattention and Hyperactivity/Impulsive subscales. The total score can range from 0 to 54 with a higher score reflecting more severe ADHD symptoms.
Time Frame: completed weekly over 8-10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adderall XR - Placebo: This is the placebo dosage week for the Adderall XR medication.
- Adderall XR - 10 mg: This is the 10 mg dosage week for the Adderall XR medication.
- Adderall XR - 20 mg: This is the 20 mg dosage week for the Adderall XR medication.
- Adderall XR - 25/30mg: This is the 25/30 mg dosage week for the Adderall XR medication.
- Focalin XR - Placebo: This is the placebo dosage week for the Focalin XR medication.
- Focalin XR - 10 mg: This is the 10 mg dosage week for the Focalin XR medication.
- Focalin XR - 20 mg: This is the 20 mg dosage week for the Focalin XR medication.
- Focalin XR - 25/30mg: This is the 25/30 mg dosage week for the Focalin XR medication.
Arm/Group | Adderall XR - Placebo | Adderall XR - 10 mg | Adderall XR - 20 mg | Adderall XR - 25/30mg | Focalin XR - Placebo | Focalin XR - 10 mg | Focalin XR - 20 mg | Focalin XR - 25/30mg
Number analyzed (Participants) | 48 | 53 | 47 | 47 | 54 | 55 | 52 | 51
units on a scale
  Inattention Symptom Subscale Scores | 16.61 (7.8) | 6.40 (8.55) | 12.2 (8.08) | 12.74 (8.38) | 17.31 (8.23) | 17.51 (7.03) | 13.33 (7.08) | 12.11 (8.72)
  Hyperactivity/Impulsivity Symptom subscale scores | 11.41 (8.55) | 10.78 (7.60) | 7.92 (6.78) | 7.67 (6.62) | 13.24 (8.91) | 10.84 (7.37) | 8.49 (7.37) | 8.49 (6.70)
  Total Symptoms scores | 28.02 (15.15) | 27.15 (14.49) | 20.12 (13.87) | 20.40 (13.68) | 30.58 (15.33) | 28.35 (12.74) | 21.82 (12.72) | 20.41 (13.61)

4. Secondary Outcome: Dopamine Active Transporter (DAT) 1 Gene Type Effects on ADHD Symptoms
Description: Three variations of the DAT 1 gene were observed, the 9/9 allele, the 9/10 allele and the 10/10 allele. The ADHD Rating Scale (ADHD-RS) and Clinical Global Impressions - Severity (CGI-S) measures were used to evaluate how the DAT 1 gene allele type altered the efficacy of the medication. The DAT 1 genotype did not predict differential response to Focalin XR or Adderall XR so the dose levels of each drug was combined to examine how the genotype interacted with the dose level. The ADHD-RS evaluates the severity of the participant's ADHD symptoms and includes two subscales: Inattention and Hyperactivity/Impulsivity. Both subscale scores range from 0 to 27 with a higher score representing more severe symptoms. The subscales are summed to calculate the total score which can range from 0 to 54. The CGI-S scale summarizes the clinician's impression of the participant's symptom severity and ranges from 1-7 with 1 representing normal (not at all ill) and 7 representing extremely ill.
Time Frame: 8-10 weeks
Population: The number of participants analyzed differs from the participant flow because some participants refused to provide a DNA sample for analysis or some participants did not have the allele type that was being observed. Of those that provided a DNA sample, 6 had the 9/9 allele on the DAT 1 gene, 15 had the 9/10 allele and 30 had the 10/10 allele.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 9/9 Allele: Placebo of Adderall XR: This is the Placebo dosage of Adderall XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 10 mg of Adderall XR: This is the 10 mg dosage of Adderall XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 20 mg Adderall XR: This is the 20 mg dosage of Adderall XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 25/30mg of Adderall XR: This is the 25/30 mg dosage of Adderall XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: Placebo of Focalin XR: This is the placebo dosage of Focalin XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 10 mg of Focalin XR: This is the 10 mg dosage of Focalin XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 20 mg of Focalin XR: This is the 20 mg dosage of Focalin XR medication phase for the participants with the 9/9 allele
- 9/9 Allele: 25/30 mg of Focalin XR: This is the 25/30 mg dosage of Focalin XR medication phase for the participants with the 9/9 allele
- 9/10 Allele: Placebo of Adderall XR: This is the Placebo dosage of Adderall XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 10 mg of Adderall XR: This is the 10 mg dosage of Adderall XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 20 mg of Adderall XR: This is the 20 mg dosage of Adderall XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 25/30 mg of Adderall XR: This is the 25/30 mg dosage of Adderall XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: Placebo of Focalin XR: This is the Placebo dosage of Focalin XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 10 mg of Focalin XR: This is the 10 mg dosage of Focalin XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 20 mg of Focalin XR: This is the 20 mg dosage of Focalin XR medication phase for the participants with the 9/10 allele
- 9/10 Allele: 25/30 mg of Focalin XR: This is the 25/30 mg dosage of Focalin XR medication phase for the participants with the 9/10 allele
- 10/10 Allele: Placebo of Adderall XR: This is the Placebo dosage of Adderall XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 10 mg of Adderall XR: This is the 10 mg dosage of Adderall XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 20 mg of Adderall XR: This is the 20 mg dosage of Adderall XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 25/30 mg of Adderall XR: This is the 25/30 mg dosage of Adderall XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: Placebo of Focalin XR: This is the Placebo dosage of Focalin XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 10 mg of Focalin XR: This is the 10 mg dosage of Focalin XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 20 mg of Focalin XR: This is the 20 mg dosage of Focalin XR medication phase for the participants with the 10/10 allele
- 10/10 Allele: 25/30mg of Focaling XR: This is the 25/30 mg dosage of Focalin XR medication phase for the participants with the 10/10 allele
Arm/Group | 9/9 Allele: Placebo of Adderall XR | 9/9 Allele: 10 mg of Adderall XR | 9/9 Allele: 20 mg Adderall XR | 9/9 Allele: 25/30mg of Adderall XR | 9/9 Allele: Placebo of Focalin XR | 9/9 Allele: 10 mg of Focalin XR | 9/9 Allele: 20 mg of Focalin XR | 9/9 Allele: 25/30 mg of Focalin XR | 9/10 Allele: Placebo of Adderall XR | 9/10 Allele: 10 mg of Adderall XR | 9/10 Allele: 20 mg of Adderall XR | 9/10 Allele: 25/30 mg of Adderall XR | 9/10 Allele: Placebo of Focalin XR | 9/10 Allele: 10 mg of Focalin XR | 9/10 Allele: 20 mg of Focalin XR | 9/10 Allele: 25/30 mg of Focalin XR | 10/10 Allele: Placebo of Adderall XR | 10/10 Allele: 10 mg of Adderall XR | 10/10 Allele: 20 mg of Adderall XR | 10/10 Allele: 25/30 mg of Adderall XR | 10/10 Allele: Placebo of Focalin XR | 10/10 Allele: 10 mg of Focalin XR | 10/10 Allele: 20 mg of Focalin XR | 10/10 Allele: 25/30mg of Focaling XR
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 3 | 5 | 4 | 4 | 14 | 15 | 14 | 14 | 13 | 15 | 12 | 10 | 30 | 30 | 29 | 26 | 27 | 27 | 27 | 26
units on a scale
  ADHD-RS Inattention subscale score | 18.60 (9.61) | 18.83 (10.59) | 19.00 (8.51) | 15.40 (9.18) | 19.33 (7.51) | 22.20 (4.76) | 16.75 (8.81) | 12.50 (9.81) | 18.64 (6.55) | 16.27 (7.33) | 15.86 (6.71) | 13.43 (7.95) | 18.08 (8.51) | 16.93 (5.59) | 13.36 (8.27) | 13.70 (9.86) | 15.07 (8.14) | 16.13 (9.35) | 9.36 (7.88) | 11.96 (8.65) | 16.44 (8.44) | 16.56 (7.92) | 12.56 (6.64) | 11.15 (8.61)
  ADHD-RS Hyperactivity/Impulsivity subscale score | 12.80 (8.90) | 18.33 (10.03) | 14.80 (8.07) | 10.40 (9.96) | 17.33 (2.52) | 17.40 (4.77) | 14.00 (9.13) | 9.00 (7.07) | 9.36 (8.95) | 10.67 (7.74) | 8.36 (7.04) | 6.43 (6.95) | 8.92 (9.38) | 8.27 (7.23) | 6.73 (7.04) | 7.00 (7.02) | 11.87 (8.76) | 9.63 (6.83) | 7.07 (6.18) | 7.50 (5.70) | 13.74 (9.19) | 10.63 (7.14) | 8.41 (6.34) | 8.65 (6.46)
  ADHD-RS total score | 31.40 (18.06) | 37.17 (20.55) | 33.80 (16.33) | 25.80 (19.03) | 36.67 (6.43) | 39.60 (8.44) | 30.75 (17.63) | 24.00 (17.19) | 28.00 (13.59) | 26.80 (13.14) | 24.21 (13.01) | 19.86 (12.84) | 27.08 (15.71) | 25.20 (11.89) | 20.09 (13.71) | 20.70 (15.84) | 26.93 (16.05) | 25.77 (14.33) | 16.43 (13.01) | 19.46 (13.20) | 30.19 (16.49) | 27.19 (12.93) | 20.96 (11.98) | 19.81 (13.26)
  CGI-S score | 4.40 (0.55) | 4.33 (1.51) | 4.80 (1.30) | 4.00 (1.58) | 4.67 (0.58) | 4.60 (0.55) | 4.50 (1.29) | 4.00 (1.63) | 4.36 (1.08) | 4.07 (1.03) | 3.71 (1.14) | 3.50 (1.40) | 4.31 (0.95) | 4.27 (0.70) | 3.58 (1.38) | 3.90 (1.66) | 4.17 (1.39) | 4.07 (1.48) | 3.21 (1.32) | 3.54 (1.24) | 4.15 (1.29) | 4.19 (0.83) | 3.52 (1.12) | 3.31 (1.26)

5. Secondary Outcome: Clinical Global Impression - Severity
Description: The CGI-S scale summarizes the clinician's impression of the participant's symptom severity and ranges from 1-7 with 1 representing normal (not at all ill) and 7 representing extremely ill.
Time Frame: 8-10 weeks
Population: The number of participants analyzed differs from the participant flow in the Focalin XR groups because the CGI-S was not completed for every participant. The same is true for the Adderall XR - 25/30mg group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adderall XR - 25/30 mg: This is the 25/30 mg dosage week for the Adderall XR medication.
- Focalin - 10 mg: This is the 10 mg dosage week for the Focalin XR medication.
- Focalin XR - 25/30 mg: This is the 25/30 mg dosage week for the Focalin XR medication.
Arm/Group | Adderall XR - Placebo | Adderall XR - 10 mg | Adderall XR - 20 mg | Adderall XR - 25/30 mg | Focalin XR - Placebo | Focalin - 10 mg | Focalin XR - 20 mg | Focalin XR - 25/30 mg
Number analyzed (Participants) | 54 | 55 | 52 | 48 | 45 | 51 | 46 | 44
units on a scale | 4.26 (1.18) | 4.09 (1.29) | 3.48 (1.34) | 3.56 (1.27) | 4.24 (1.13) | 4.24 (0.76) | 3.63 (1.20) | 3.55 (1.35)

6. Secondary Outcome: Weiss Functional Impairment Rating Scale (WFIRS)
Description: The WFIRS consists of 50 questions where respondents are asked to rate their child's functional impairment. The items of the WFIRS are scored on a four point Likert-type rating scale: 0 (never or not at all), 1 (sometimes or somewhat), 2 (often or much) or 3 (very often or very much) and aggregated to produce six domain scores: Family (ranges between 0-24), Learning or School (ranges between 0-33), Self-Concept (ranges between 0-15), Social Activities (ranges between 0-27), Life Skills (ranges between 0-36), and Risky Activities (ranges between 0-42). The subscales are scored by summing the responses in the subsection. The Total score is the sum of all the responses and it ranges between 0-150. The higher the score in each of the subscales the more impairment is recorded, this is also true for the total score.
Time Frame: 8-10 weeks
Population: The number of participants analyzed differs from the participant flow in all of the groups besides the Adderall XR - 10mg group because the WFIRS was not completed for every participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adderall XR - Placebo | Adderall XR - 10 mg | Adderall XR - 20 mg | Adderall XR - 25/30mg | Focalin XR - Placebo | Focalin XR - 10 mg | Focalin XR - 20 mg | Focalin XR - 25/30mg
Number analyzed (Participants) | 53 | 55 | 51 | 47 | 44 | 48 | 46 | 42
units on a scale
  Family subscale score | 6.72 (6.13) | 7.02 (6.41) | 6.35 (6.10) | 6.70 (7.14) | 7.39 (7.14) | 7.35 (6.09) | 6.50 (6.42) | 6.50 (6.46)
  Learning subscale score | 6.74 (5.63) | 8.75 (6.70) | 6.86 (6.19) | 6.21 (5.62) | 9.30 (6.34) | 9.25 (5.94) | 7.54 (5.24) | 7.39 (5.78)
  Life skills subscale score | 7.43 (4.32) | 7.91 (4.78) | 7.44 (4.99) | 7.34 (4.45) | 8.30 (4.76) | 7.65 (4.44) | 8.30 (5.48) | 7.60 (5.66)
  Self-concept subscale score | 1.11 (1.46) | 1.59 (2.05) | 1.42 (1.80) | 1.06 (1.61) | 1.25 (1.97) | 1.19 (1.47) | 1.33 (1.61) | 1.31 (1.97)
  Social activities subscale score | 3.51 (3.53) | 3.91 (3.81) | 2.98 (3.10) | 3.06 (4.05) | 3.73 (4.14) | 3.85 (3.57) | 3.54 (3.40) | 3.17 (3.98)
  Risky activities subscale score | 2.19 (2.56) | 1.94 (2.30) | 2.24 (3.41) | 1.68 (2.23) | 1.91 (1.64) | 1.96 (2.12) | 1.78 (1.78) | 1.67 (1.73)
  Total score | 27.70 (17.03) | 31.06 (18.93) | 27.32 (19.53) | 26.23 (19.74) | 20.91 (17.50) | 31.13 (17.11) | 29.20 (17.71) | 27.45 (18.54)

ADVERSE EVENTS:
Time Frame: 8-10 weeks. Adverse events were collected from participants while they were in the study, this time frame ranged from 8-10 weeks.
Description: At each weekly visit, children and their parents met with the investigators and research staff. Parents completed the Stimulant Side Effects Rating scale (SERS), a 17-item scale that is rated on a 10-point (0-9) scale ranging from absent to serious.
Groups:
- Placebo of Focalin XR: Each participant recieved placebo of Focalin XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 10mg of Focalin XR: Each participant recieved 10 mg of Focalin XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 20 mg of Focalin XR: Each participant recieved 20 mg of Focalin XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 25/30mg of Focalin XR: Each participant recieved 25/30 mg (depending on weight) of Focalin XR once during the first four weeks or last four weeks depending on the randomization schedule.
- Placebo of Adderall XR: Each participant recieved placebo of Adderall XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 10mg of Adderall XR: Each participant recieved 10 mg of Adderall XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 20 mg of Adderall XR: Each participant recieved 20 mg of Adderall XR once during the first four weeks or last four weeks depending on the randomization schedule.
- 25/30mg of Adderall XR: Each participant recieved 25/30 mg of Adderall XR once during the first four weeks or last four weeks depending on the randomization schedule.
Arm/Group | Placebo of Focalin XR | 10mg of Focalin XR | 20 mg of Focalin XR | 25/30mg of Focalin XR | Placebo of Adderall XR | 10mg of Adderall XR | 20 mg of Adderall XR | 25/30mg of Adderall XR
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/53 | 1/47 | 0/47 | 0/54 | 0/55 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 16/48 | 23/53 | 32/47 | 22/47 | 23/54 | 35/55 | 29/52 | 31/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo of Focalin XR (N=48) | 10mg of Focalin XR (N=53) | 20 mg of Focalin XR (N=47) | 25/30mg of Focalin XR (N=47) | Placebo of Adderall XR (N=54) | 10mg of Adderall XR (N=55) | 20 mg of Adderall XR (N=52) | 25/30mg of Adderall XR (N=51)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject shaking in bed,unresponsive,eyes rolled upward. Taken to ER. ECG showed possible prolonged QTc. Subject evaluated overnight. No other events. Diagnosed on 12/29 with "benign rolandic seizures." No further cardiac evaluation recommended.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo of Focalin XR (N=48) | 10mg of Focalin XR (N=53) | 20 mg of Focalin XR (N=47) | 25/30mg of Focalin XR (N=47) | Placebo of Adderall XR (N=54) | 10mg of Adderall XR (N=55) | 20 mg of Adderall XR (N=52) | 25/30mg of Adderall XR (N=51)
Insomnia or trouble sleeping (Psychiatric disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3) | 3 (3) | 7 (7) | 6 (6) | 4 (4)
Talk less (General disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Loss of Appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 6 (6) | 3 (3) | 2 (2) | 5 (5) | 7 (7) | 6 (6)
Irritable (General disorders) | 3 (3) | 1 (1) | 7 (7) | 5 (5) | 3 (3) | 4 (4) | 5 (5) | 1 (1)
Stomach Ache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Headache (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Nail biting (General disorders) | 3 (3) | 7 (7) | 9 (9) | 6 (6) | 4 (4) | 9 (9) | 7 (7) | 5 (5)
Euphoric (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nightmare (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stares (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Uninterested (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sadness (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Crying (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tics (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early withdrawal or loss of contact during the study, the sample size for analysis was smaller.

The dosing design of the study may have led to more adverse events than would occur in clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No